CLINICAL TRIAL: NCT02319681
Title: Reminiscence, Anxiety and Early Alzheimer's Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI relocated to UNCP; Study is not being transferred
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, William Puentes, Clinical Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00075912
Record Dates: First submitted 2014-12-15; First posted 2014-12-18 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Alzheimer's Disease
Keywords: Caregivers; Anxiety; Depression
MeSH Terms: conditions — Alzheimer Disease; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simple Reminiscence (SR) caregiver (Experimental): Subjects are caregivers for a persons with EAD and will be administered SR intervention and an attention control treatment four times
  Interventions: Behavioral: Simple Reminiscence (SR); Behavioral: Attention Control (AC)
- Simple Reminiscence (SR) EAD (Experimental): Subjects are persons with EAD and will be administered SR intervention and an attention control treatment four times
  Interventions: Behavioral: Simple Reminiscence (SR); Behavioral: Attention Control (AC)

INTERVENTIONS:
Behavioral: Simple Reminiscence (SR) — SR is a 30-minute psychoeducational activity administered by a trained RA at 4 home visits (week 2, week 3, week 7, and week 19). SR has a didactic component using the SR manual that the couple retains, viewing one of the brief video-vignettes illustrating the application of reminiscence techniques (a different video-vignette will be viewed at each visit), and facilitation of caregiver practice in applying the techniques, using a recent example of anxiety-linked experience of the person with EAD.
Behavioral: Attention Control (AC) — AC is a 30-minute in which the person with EAD, the caregiver and the RA review and discuss the day's newspaper headlines. The RA will use communication techniques specifically designed to keep the conversation present focused at 4 home visits (week 2, week 3, week 7, and week 19).

SUMMARY:
This study seeks to establish the acceptability and evaluate the limited efficacy of Simple Reminiscence (SR), a home-delivered non-pharmacological intervention designed to relieve stress, improve affect, and prevent or quell disruptive or maladaptive behaviors in community-residing individuals diagnosed with early Alzheimer's disease (EAD). Unmanaged episodes of anxiety can be antecedents of maladaptive behaviors, including agitation, anger, and sometimes even violence.

SR is a dyadic strategy; both the person with EAD and the caregiver engaged the patient's memory to interrupt a current episode of anxiety.

DETAILED DESCRIPTION:
Through the intervention, family caregivers are trained to collaborate with and guide patients to access positive memories as a way to manage or move past the anxiety that plagues individuals with EAD - often arising when confronted by common complex tasks they previously were able to perform.

During the project's first six months (phase 1), the investigators will develop a series of 4 video-vignettes illustrating dyads (including one member with EAD) managing a variety of anxiety provoking scenarios associated with EAD (e.g., trouble reconciling a checkbook) through the use of SR.

During the second phase of the project, a research assistant will administer SR at four home visits. The SR intervention has three components:

1. A didactic component using the SR manual that the couple retains (15 minutes);
2. Viewing one of the brief video-vignettes illustrating the application of reminiscence techniques (5 minutes; a different video-vignette will be viewed at each visit; and
3. Facilitation of caregiver practice in applying the techniques, using a recent example of anxiety-linked experience of the person with EAD (10 minutes). The caregiver is encouraged to learn and practice the techniques in order to cue and coach the person with EAD in their use.

The attention control treatment, a Social Visit, is a 30-minute activity in which the person with EAD, the caregiver and the research assistant (RA) review and discuss the day's newspaper headlines. The RA will use communication techniques specifically designed to keep the conversation present focused.

Both members of the dyad will collect saliva to evaluate diurnal cortisol secretion.

ELIGIBILITY:
Inclusion Criteria:

* Live in the community
* Reside with a primary caregiver who must be willing to participate in all study activities (the primary caregiver must have a familial or marital relationship with the person with EAD of sufficient length to support reminiscence activity [i.e., an adult child, a long-term spouse or committed partner])
* Have received a diagnosis of Early Alzheimer's Disease from a primary care provider
* Achieve a score on the mini-mental state examination (MMSE) between 19 and 25

Exclusion Criteria:

* Unable to give consent
* MMSE score lower than 19 or greater than 25.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Acceptability of SR and AC | Week 20
  Taped interview with the dyad will occur asking how acceptable the format, duration, and frequency of the program

SECONDARY OUTCOMES:
Number of times AC was used | Week 20
  Taped interview with the dyad will occur asking how frequently AC was used
Number of times SR was used | Week 20
  Taped interview with the dyad will occur asking how frequently SR was used
Change in Beck Depression Inventory-II (BDI-II) scale | Baseline, week 20
  BDI-II is a 21-item, self-administered tool used to measure depressive symptoms. Scores range from 0 - 63, with higher scores indicating more severe depressive symptoms.
Change in State-Trait Anxiety Inventory (STAI) scale | Baseline, week 20
  STAI is a 20-item tool that measures current anxiety symptoms with scores that range from 20 to 80, with higher scores indicating greater levels of anxiety.
Change in Katz Instrumental Activities of Daily Living (IADL) scale | Baseline, week 20
  IADL is a six-item tool assessing the degree of independence vs. dependence in basic activities of daily living, with higher scores indicating greater levels of daily functioning.
Change in Well-Being Picture Scale (WBPS) scale | Baseline, week 20
  WBPS is a 10-item non-language based pictorial scale that measures general well-being. Individuals are asked to mark the point along each scale to indicate which image they feel most like (drawings depicting a sense of high or low well-being are arranged at opposite ends of a scale).
Change in Short Psychological Well-Being Scale (SPWBS) scale | Baseline, week 20
  SPWBS is a 84-item self-report, Likert-type inventory that measures well-being across six dimensions: Self-Acceptance, Positive Relations With Others, Autonomy, Environmental Mastery, Purpose in Life, and Personal Growth. A higher score indicated a greater sense of well-being.
Change in Revised Memory and Behavior Problems Checklist (RMBPC) scale | Baseline, week 20
  RMBPC is a 24-item Likert-type caregiver-report measure of observable behavioral problems in dementia.
Caregiver's mastery of SR intervention technique | Week 20
  Simple Reminiscence Intervention Mastery Assessment (SRIMA) evaluation rubric to be used to determine the person with EAD's and their caregiver's mastery of the SR Intervention techniques.
Change in levels of cortisol | Baseline, Week 20
  Both members of the dyad will collect saliva to evaluate diurnal cortisol secretion by standard enzyme-linked immunoabsorbant assay ( ELISA).

CONTACTS AND LOCATIONS:
Overall Officials: William Puentes, PhD RN FAAN, Principal Investigator — Emory University
Locations (1):
- Emory Alzheimer's Disease Research Center, Atlanta, Georgia, United States